CLINICAL TRIAL: NCT01999400
Title: Correlation of Mesalamine Pharmacokinetics With Local Availability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Duxin Sun, Professor, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: FDA-SOL-1120920; HHSF223201300460A (Other Grant/Funding Number: U.S. Food and Drug Administration); HHSF223201000082C (Other Grant/Funding Number: U.S. Food and Drug Administration)
Record Dates: First submitted 2013-11-25; First posted 2013-12-03 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Local Drug Concentration in Gastrointestinal Tract
MeSH Terms: interventions — Mesalamine; Water

ARMS (6):
- Arm 1: Pentasa then Delzicol then Apriso then Lialda (Experimental): 1. Pentasa 500 mg capsule x 2 with 240 mL water, single dose.
  2. Washout period of 10 days.
  3. Delzicol 100 mg mesalamine x 1 with 245 mL water, single dose.
  4. Washout period of 10 days.
  5. Apriso 375 mg capsule x 3 with 240 mL water, single dose.
  6. Washout period of 10 days.
  7. Lialda 1200 mg tablet x 1 with 240 mL water, single dose.
  Interventions: Drug: Pentasa 500 mg capsule x 2 with 240 mL water; single dose; Drug: Apriso 375 mg capsule x 3 with 240 mL water; single dose; Drug: Lialda 1200 mg tablet x 1 with 240 mL water; single dose; Drug: Delzicol 100 mg mesalamine x 1 with 245 mL water; single dose
- Arm 2: Pentasa then Delzicol then Lialda then Apriso (Experimental): 1. Pentasa 500 mg capsule x 2 with 240 mL water, single dose.
  2. Washout period of 10 days.
  3. Delzicol 100 mg mesalamine x 1 with 245 mL water, single dose.
  4. Washout period of 10 days.
  5. Lialda 1200 mg tablet x 1 with 240 mL water, single dose.
  6. Washout period of 10 days.
  7. Apriso 375 mg capsule x 3 with 240 mL water, single dose.
  Interventions: Drug: Pentasa 500 mg capsule x 2 with 240 mL water; single dose; Drug: Apriso 375 mg capsule x 3 with 240 mL water; single dose; Drug: Lialda 1200 mg tablet x 1 with 240 mL water; single dose; Drug: Delzicol 100 mg mesalamine x 1 with 245 mL water; single dose
- Arm 3: Apriso then Delzicol then Pentasa then Lialda (Experimental): 1. Apriso 375 mg capsule x 3 with 240 mL water, single dose.
  2. Washout period of 10 days.
  3. Delzicol 100 mg mesalamine x 1 with 245 mL water, single dose.
  4. Washout period of 10 days.
  5. Pentasa 500 mg capsule x 2 with 240 mL water, single dose.
  6. Washout period of 10 days.
  7. Lialda 1200 mg tablet x 1 with 240 mL water, single dose.
  Interventions: Drug: Pentasa 500 mg capsule x 2 with 240 mL water; single dose; Drug: Apriso 375 mg capsule x 3 with 240 mL water; single dose; Drug: Lialda 1200 mg tablet x 1 with 240 mL water; single dose; Drug: Delzicol 100 mg mesalamine x 1 with 245 mL water; single dose
- Arm 4: Apriso then Delzicol then Lialda then Pentasa (Experimental): 1. Apriso 375 mg capsule x 3 with 240 mL water, single dose.
  2. Washout period of 10 days.
  3. Delzicol 100 mg mesalamine x 1 with 245 mL water, single dose.
  4. Washout period of 10 days.
  5. Lialda 1200 mg tablet x 1 with 240 mL water, single dose.
  6. Washout period of 10 days.
  7. Pentasa 500 mg capsule x 2 with 240 mL water, single dose.
  Interventions: Drug: Pentasa 500 mg capsule x 2 with 240 mL water; single dose; Drug: Apriso 375 mg capsule x 3 with 240 mL water; single dose; Drug: Lialda 1200 mg tablet x 1 with 240 mL water; single dose; Drug: Delzicol 100 mg mesalamine x 1 with 245 mL water; single dose
- Arm 5: Lialda then Delzicol then Pentasa then Apriso (Experimental): 1. Lialda 1200 mg tablet x 1 with 240 mL water, single dose.
  2. Washout period of 10 days.
  3. Delzicol 100 mg mesalamine x 1 with 245 mL water, single dose.
  4. Washout period of 10 days.
  5. Pentasa 500 mg capsule x 2 with 240 mL water, single dose.
  6. Washout period of 10 days.
  7. Apriso 375 mg capsule x 3 with 240 mL water, single dose.
  Interventions: Drug: Pentasa 500 mg capsule x 2 with 240 mL water; single dose; Drug: Apriso 375 mg capsule x 3 with 240 mL water; single dose; Drug: Lialda 1200 mg tablet x 1 with 240 mL water; single dose; Drug: Delzicol 100 mg mesalamine x 1 with 245 mL water; single dose
- Arm 6: Lialda then Delzicol then Apriso then Pentasa (Experimental): 1. Lialda 1200 mg tablet x 1 with 240 mL water, single dose.
  2. Washout period of 10 days.
  3. Delzicol 100 mg mesalamine x 1 with 245 mL water, single dose.
  4. Washout period of 10 days.
  5. Apriso 375 mg capsule x 3 with 240 mL water, single dose.
  6. Washout period of 10 days.
  7. Pentasa 500 mg capsule x 2 with 240 mL water, single dose.
  Interventions: Drug: Pentasa 500 mg capsule x 2 with 240 mL water; single dose; Drug: Apriso 375 mg capsule x 3 with 240 mL water; single dose; Drug: Lialda 1200 mg tablet x 1 with 240 mL water; single dose; Drug: Delzicol 100 mg mesalamine x 1 with 245 mL water; single dose

INTERVENTIONS:
Drug: Pentasa 500 mg capsule x 2 with 240 mL water; single dose
Drug: Apriso 375 mg capsule x 3 with 240 mL water; single dose
Drug: Lialda 1200 mg tablet x 1 with 240 mL water; single dose
Drug: Delzicol 100 mg mesalamine x 1 with 245 mL water; single dose

SUMMARY:
This study is designed to provide data to the FDA correlating pharmacokinetics with local availability of medications within the gastrointestinal tract. This study will support the establishment of scientifically based standards for evaluating drugs which act locally within the gastrointestinal tract. Specific objectives of this study are to: (1) quantify how the plasma concentrations of mesalamine, an agent used to treat inflammatory bowel disease, are correlated with the concentrations in gastrointestinal fluids; and (2) improve the physiologically based models for drug absorption from the intestine. Information from this study in concert with in vitro dissolution data will be used to evaluate in vivo-in vitro correlation (IVIVC) for concentrations in plasma and intestinal lumen and dissolution of mesalamine products.

DETAILED DESCRIPTION:
This study evaluated the pharmacokinetics of mesalamine and its major metabolite of mesalamine known as N-acetyl-mesalamine in plasma. Mesalamine is available in different formulations that control the rate at which they are released in the gastrointestinal tract. Three formulations of mesalamine, Pentasa, Apriso, and Lialda, were studied in the crossover phase, while an oral solution formulation of mesalamine was studied in the single-arm phase. Each subject participated in a crossover phase study with one of the three formulations assigned at random using block randomization. Then the subject entered the single-arm phase study. After participation in one crossover phase study and one single-arm phase study, the subject could opt to participate in crossover phase studies using the other formulations also chosen at random until all three formulations were studied. The single-arm phase study was not repeated on returning subjects who participated in more than one crossover phase study.

ELIGIBILITY:
Inclusion Criteria

1. Adults age 18 to 55.
2. Male or female voluntarily able to give informed consent.
3. Body mass index (BMI) 18.5 to 35.

Exclusion Criteria

1. Adults unable to consent for themselves or mentally incapacitated.
2. Prisoners.
3. Significant clinical illness within 3 weeks prior to Screening.
4. Use of concomitant medications within 2 weeks prior to receiving study drug, including but not limited to prescription drugs, herbal and dietary supplements, over the counter medications, and vitamins. Oral contraception is permitted.
5. History of gastrointestinal surgery.
6. History of allergy to non-steroidal anti-inflammatory drugs (NSAIDs) or to any of the ingredients of Asacol, Pentasa, Apriso, or Lialda.
7. History of severe allergic diseases including drug allergies, with the exception of seasonal allergies.
8. Any other factor, condition, or disease, including, but not limited to, cardiovascular, renal, hepatic, or gastrointestinal disorders that may, in the opinion of the Investigator, jeopardize the safety of the patient or impact the validity of the study results.
9. History of drug addiction or alcohol abuse within the past 12 months.
10. Pregnant or lactating females.
11. Surgery within the past 3 months.
12. Received an investigational drug within 60 days prior to receiving the study drug.
13. Any clinically significant abnormal lab values during Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-04; Primary Completion 2015-09 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Duxin Sun, Ph.D., Principal Investigator — University of Michigan, College of Pharmacy
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Lionberger RA. FDA critical path initiatives: opportunities for generic drug development. AAPS J. 2008;10(1):103-9. doi: 10.1208/s12248-008-9010-2. Epub 2008 Feb 20. PMID 18446510

RESULTS

PARTICIPANT FLOW:
Period: First Intervention (1 Day)
Arm/Group | Arm 1: Pentasa Then Delzicol Then Apriso Then Lialda | Arm 2: Pentasa Then Delzicol Then Lialda Then Apriso | Arm 3: Apriso Then Delzicol Then Pentasa Then Lialda | Arm 4: Apriso Then Delzicol Then Lialda Then Pentasa | Arm 5: Lialda Then Delzicol Then Pentasa Then Apriso | Arm 6: Lialda Then Delzicol Then Apriso Then Pentasa
Started | 6 | 6 | 5 | 5 | 4 | 4
Completed | 4 | 4 | 3 | 2 | 4 | 3
Not Completed | 2 | 2 | 2 | 3 | 0 | 1
Period: Washout (10 Days)
Arm/Group | Arm 1: Pentasa Then Delzicol Then Apriso Then Lialda | Arm 2: Pentasa Then Delzicol Then Lialda Then Apriso | Arm 3: Apriso Then Delzicol Then Pentasa Then Lialda | Arm 4: Apriso Then Delzicol Then Lialda Then Pentasa | Arm 5: Lialda Then Delzicol Then Pentasa Then Apriso | Arm 6: Lialda Then Delzicol Then Apriso Then Pentasa
Started | 5 | 4 | 3 | 2 | 3 | 3
Completed | 5 | 4 | 3 | 2 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | Arm 1: Pentasa Then Delzicol Then Apriso Then Lialda | Arm 2: Pentasa Then Delzicol Then Lialda Then Apriso | Arm 3: Apriso Then Delzicol Then Pentasa Then Lialda | Arm 4: Apriso Then Delzicol Then Lialda Then Pentasa | Arm 5: Lialda Then Delzicol Then Pentasa Then Apriso | Arm 6: Lialda Then Delzicol Then Apriso Then Pentasa
Started | 5 | 4 | 3 | 2 | 3 | 3
Completed | 5 | 4 | 3 | 2 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (10 Days)
Arm/Group | Arm 1: Pentasa Then Delzicol Then Apriso Then Lialda | Arm 2: Pentasa Then Delzicol Then Lialda Then Apriso | Arm 3: Apriso Then Delzicol Then Pentasa Then Lialda | Arm 4: Apriso Then Delzicol Then Lialda Then Pentasa | Arm 5: Lialda Then Delzicol Then Pentasa Then Apriso | Arm 6: Lialda Then Delzicol Then Apriso Then Pentasa
Started | 2 | 0 | 1 | 1 | 1 | 1
Completed | 2 | 0 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention (1 Day)
Arm/Group | Arm 1: Pentasa Then Delzicol Then Apriso Then Lialda | Arm 2: Pentasa Then Delzicol Then Lialda Then Apriso | Arm 3: Apriso Then Delzicol Then Pentasa Then Lialda | Arm 4: Apriso Then Delzicol Then Lialda Then Pentasa | Arm 5: Lialda Then Delzicol Then Pentasa Then Apriso | Arm 6: Lialda Then Delzicol Then Apriso Then Pentasa
Started | 2 | 0 | 1 | 1 | 1 | 1
Completed | 2 | 0 | 1 | 1 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Period: Washout (10 Days)
Arm/Group | Arm 1: Pentasa Then Delzicol Then Apriso Then Lialda | Arm 2: Pentasa Then Delzicol Then Lialda Then Apriso | Arm 3: Apriso Then Delzicol Then Pentasa Then Lialda | Arm 4: Apriso Then Delzicol Then Lialda Then Pentasa | Arm 5: Lialda Then Delzicol Then Pentasa Then Apriso | Arm 6: Lialda Then Delzicol Then Apriso Then Pentasa
Started | 1 | 0 | 1 | 0 | 0 | 0
Completed | 1 | 0 | 1 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Fourth Intervention (1 Day)
Arm/Group | Arm 1: Pentasa Then Delzicol Then Apriso Then Lialda | Arm 2: Pentasa Then Delzicol Then Lialda Then Apriso | Arm 3: Apriso Then Delzicol Then Pentasa Then Lialda | Arm 4: Apriso Then Delzicol Then Lialda Then Pentasa | Arm 5: Lialda Then Delzicol Then Pentasa Then Apriso | Arm 6: Lialda Then Delzicol Then Apriso Then Pentasa
Started | 1 | 0 | 1 | 0 | 0 | 0
Completed | 1 | 0 | 1 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants who were randomized to one of the six arms of this study:
  Arm 1: Pentasa then Delzicol then Apriso then Lialda Arm 2: Pentasa then Delzicol then Lialda then Apriso Arm 3: Apriso then Delzicol then Pentasa then Lialda Arm 4: Apriso then Delzicol then Lialda then Pentasa Arm 5: Lialda then Delzicol then Pentasa then Apriso Arm 6: Lialda then Delzicol then Apriso then Pentasa
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.9 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 21
Body Mass Index [Mean (Standard Deviation); unit: kg per m squared] | 26.9 (5.6)

OUTCOME MEASURES:

1. Primary Outcome: The AUC of Mesalamine in Plasma
Description: The AUC is the area under the concentration-time curve from time 0 to last time point. The data are organized by the different drug formulations of mesalamine, which include Pentasa (0 to 72 hours), Apriso (0 to 72 hours), Lialda (0 to 96 hours), and Delzicol (0 to 24 hours). The AUC is measured in units of nanomoles of mesalamine per liter of plasma (nM) multiplied by time in hours (nM*h). The AUC results are reported over the time-period because this provides a more meaningful comparison of potential differences in the bioequivalence of formulations.
Time Frame: 0 hours pre-dose and up to 96 hours post-dose
Measure: Mean (Standard Deviation); unit: nM*h
Groups:
- Pentasa: Pentasa 500 mg capsule x 2 with 240 mL water, single dose
  Pentasa 500 mg capsule x 2 with 240 mL water; single dose
- Apriso: Apriso 375 mg capsule x 3 with 240 mL water, single dose
  Apriso 375 mg capsule x 3 with 240 mL water; single dose
- Lialda: Lialda 1200 mg tablet x 1 with 240 mL water, single dose
  Lialda 1200 mg tablet x 1 with 240 mL water; single dose
- Delzicol: Delzicol 100 mg mesalamine x 1 with 245 mL water, single dose
  Delzicol 100 mg mesalamine x 1 with 245 mL water; single dose
Arm/Group | Pentasa | Apriso | Lialda | Delzicol
Number analyzed (Participants) | 10 | 7 | 9 | 20
nM*h | 40.8 (29.5) | 57.6 (24.1) | 36.8 (16.0) | 7.9 (3.7)

2. Primary Outcome: The AUC of Metabolite (N-acetyl-mesalamine) in Plasma
Description: The AUC is the area under the concentration-time curve from time 0 to last time point. The data are organized by the different drug formulations of mesalamine, which include Pentasa (0 to 72 hours), Apriso (0 to 72 hours), Lialda (0 to 96 hours), and Delzicol (0 to 24 hours). The AUC is measured in units of nanomoles of N-acetyl-mesalamine per liter of plasma (nM) multiplied by time in hours (nM*h). The AUC results are reported over the time-period because this provides a more meaningful comparison of potential differences in the bioequivalence of formulations.
Time Frame: 0 hours pre-dose and up to 96 hours post-dose
Measure: Mean (Standard Deviation); unit: nM*h
Arm/Group | Pentasa | Apriso | Lialda | Delzicol
Number analyzed (Participants) | 10 | 7 | 9 | 20
nM*h | 162 (59.7) | 189 (92.2) | 124 (80.5) | 20.4 (7.7)

3. Secondary Outcome: The AUC of Mesalamine in Distal Jejunum
Description: The AUC is the area under the concentration-time curve from time 0 to 7 hours. The data are organized by the different drug formulations of mesalamine, which include Pentasa, Apriso, and Lialda. The AUC is measured in units of micromoles of mesalamine per liter of plasma (µM) multiplied by time in hours (µM*h).The AUC results are reported over the time-period because this provides a more meaningful comparison of potential differences in the bioequivalence of formulations. The solution formulation (Delzicol) was not administered in this portion of the study. Therefore no results pertaining to the solution formulation are included in this outcome measure.
Time Frame: 0 hours pre-dose and up to 7 hours post-dose
Population: The number of subjects that were administered Pentasa, Apriso, Lialda were 10, 7, and 9, respectively. However, we were only able to collect gastrointestinal fluid from the distal jejunum for only 3 subjects in each of these arms due to the placement of the gastrointestinal tube.
Measure: Mean (Standard Deviation); unit: uM*h
Arm/Group | Pentasa | Apriso | Lialda
Number analyzed (Participants) | 3 | 3 | 3
uM*h | 8456 (7444) | 4923 (8506) | 2.9 (3.9)

4. Secondary Outcome: The AUC of Metabolite (N-acetyl-mesalamine) in Distal Jejunum
Description: as for outcome 3
Time Frame: 0 hours pre-dose and up to 7 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: uM*h
Arm/Group | Pentasa | Apriso | Lialda
Number analyzed (Participants) | 3 | 3 | 3
uM*h | 5048 (5553) | 1225 (2024) | 3.4 (3.4)

ADVERSE EVENTS:
Arm/Group | Pentasa | Apriso | Lialda | Delzicol
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13 | 0/11 | 0/20
Other Adverse Events (participants affected / at risk) | 0/14 | 0/13 | 1/11 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pentasa (N=14) | Apriso (N=13) | Lialda (N=11) | Delzicol (N=20)
vasovagal syncope (Nervous system disorders) | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Evaluation of healthy volunteers that may not reflect patients with inflammatory bowel disease.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No